CLINICAL TRIAL: NCT01227486
Title: Verification of Endotracheal Tube Placement by Ultrasound in the Obese Patient
Status: Completed | Type: Observational
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Carsten Boe Pedersen, Department of Anaesthesiology, Copenhagen University Hospital Bispebjerg
Other Study IDs: disb-01-10
Record Dates: First submitted 2010-10-20; First posted 2010-10-25 (Estimated); Last update posted 2010-11-24 (Estimated); Status verified 2010-11

CONDITIONS: Intubation, Intratracheal; Obesity
Keywords: Intubation, intratracheal; Ultrasonography; Auscultation; Capnography; Obesity
MeSH Terms: conditions — Obesity | interventions — Ultrasonography

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Obese patients for planned surgery and endotracheal intubation
  Interventions: Device: Ultrasound

INTERVENTIONS:
Device: Ultrasound — Ultrasound scan just proximal to the suprasternal notch during intubation and ultrasound scan of both lungs during ventilation

SUMMARY:
The purpose of this study is to determine whether verification of correct tube placement after endotracheal intubation in the obese patient can be conducted as fast with ultrasound as with the conventional method of combined auscultation and capnography.

The investigators hypothesize that ultrasound is a faster method for verifying correct endotracheal tube placement in the obese patient than combined auscultation and capnography.

DETAILED DESCRIPTION:
Both verification methods are conducted in all patients and patients act as their own control

ELIGIBILITY:
Inclusion Criteria:

* Planned for bariatric surgery in general anaesthesia
* Planned for endotracheal intubation
* BMI above 30

Exclusion Criteria:

* Predicted difficult airway in the pre-anaesthesia airway evaluation.
* Unpredicted difficult airway during induction of anaesthesia where assistance is needed by the investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Obese patients admitted for planned bariatric surgery on Glostrup Hospital, Denmark
Sampling Method: Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2010-10

PRIMARY OUTCOMES:
Difference in time to correct verification of endotracheal tube placement between ultrasound and combined auscultation and capnography | 0 to 1 hour

SECONDARY OUTCOMES:
Difference in time to correct verification of endotracheal tube placement between ultrasound and auscultation alone | 0 to 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Dan Isbye, M.D., PhD., Principal Investigator — Department of Anaesthesiology, Copenhagen University Hospital Bispbjerg
Locations (1):
- Department of Anaesthesiology, Bariatric section. Copenhagen University Hospital Glostrup, Glostrup Municipality, Denmark